CLINICAL TRIAL: NCT05252780
Title: "My Body, My Rhythm, My Voice": a Community Dance Intervention Engaging Breast Cancer Survivors in Physical Activity in a Middle-income Country
Brief Title: A Community Dance Intervention Engaging Breast Cancer Survivors in a Middle-income Country
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olga Lucia Sarmiento (Other)
Collaborators: Stanford University (Other); Universidad Manuela Beltrán (Other); Pontificia Universidad Javeriana (Other); Hospital de San Jose (Other); University of California, Los Angeles (Other); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Olga Lucia Sarmiento, Professor School of Medicine, Epidemiology, Universidad de los Andes, Bogota, Colombia, University of Los Andes, Columbia
Organization: University of Los Andes, Columbia (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P20CA217199-9492018; P20CA217199 (NIH)
Record Dates: First submitted 2021-12-07; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Physical Inactivity; Breast Cancer
Keywords: Breast cancer survivors; Physical activity; Behavior change intervention; Community-based program; Mixed-methods assessment; Middle-income setting
MeSH Terms: conditions — Sedentary Behavior; Breast Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): My Body, My Rhythm, My Voice
  Interventions: Behavioral: My Body, My Rhythm, My Voice
- Control group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: My Body, My Rhythm, My Voice — My Body was a behavioral intervention informed by the social cognitive and self-determination theories. Based on the discussions and a systematic review of the literature, we designed the 8-week, 3 times/week rumba physical activity intervention. The goal of the intervention was to gradually increase all participants' physical activity levels to achieve significant health benefits. As part of the physical activity intervention, participants were also taught by their instructor during each class how to utilize behavioral and cognitive self-regulatory skills to increase and maintain their physical activity participation. Examples of such skills were action planning, coping planning, counter conditioning, self-evaluation, among others.
  Other Names: My Body
  Arms: Intervention group

SUMMARY:
Interventions to promote physical activity among women breast cancer survivors (BCS) in low to middle-income countries are limited. We conducted a study to assess the acceptability and preliminary effectiveness of an 8-week, 3 times/week group dance intervention for BCS delivered in Bogotá, Colombia. The effect of the intervention on participants' physical activity levels, motivation to engage in physical activity, and quality of life were evaluated, and interviews were thematically analyzed to assess program acceptability.

DETAILED DESCRIPTION:
This is a quasi-experimental study with a control group and an intervention group.

The study population are patients over 18 years of age with a diagnosis of breast cancer who have received management and are currently in remission phase (more than 1 year after finishing management with chemotherapy and radiotherapy) and who do not report having any medical contraindication for the practice of physical activity (angina, acute myocardial infarction, pulmonary embolism, arterial hypertension and uncontrolled diabetes mellitus, severe lymphedema). The control group will be patients who attend their medical check-ups at the National Cancer Institute of Colombia and the intervention group will be patients who are cared for by units of the Bogotá's medical service. It will have the written approval of the ethics committee of the respective hospitals.

Being an exploratory study that investigates the acceptability and main motivations for attending physical activity sessions on a regular basis, it is considered that a sample of 30 people in the control group and 30 people in the intervention group could provide the necessary information to have in mind to develop studies with more significant sample sizes in the future.

For 8 weeks the intervention group will be offered 24 classes of musicalized directed physical activity (through a training protocol adapted for patients with this underlying pathology), and 8 craft workshops, to be held in the same space as the physical activity sessions. Additionally, at the same time, healthy habits will be promoted with the control group through text messages during 8 weeks, with a two workshops (at the beginning and the end of this period). The classes and workshops will be held at the facilities of the health provider institution in a place that guarantees the privacy of the participants.

For the recruitment of patients in the intervention group, women who were diagnosed with altered BI-RADS will be contacted by telephone. For the recruitment of patients from the control group, the head nurse who coordinates the follow-up program for breast cancer patients will be asked to invite the women in the study to participate. Additionally, all invited patients will receive the information through an attached information sheet.

Before the start of the intervention and after it, the following measurements will be made:

1. The questionnaires include questions about sociodemographic data, medical information, quality of life, general state of health, optimism and pessimism about life, anxiety and depression, perception of fatigue, knowledge about physical activity, self-efficacy in physical activity and social support for the practice of physical activity. These questionnaires will be administered by pollsters trained and registered through the Qualtrics application. These questionnaires will be applied by trained interviewers in a personal meeting in both health centers, in a space that ensures the confidentiality and security of the information.
2. Objective measurements that include levels of physical activity by accelerometry and body composition by bio-impedance. These measurements will be carried out by a professional in Respiratory Therapy in the facilities of the institution that provides services where the women have been recruited, as appropriate control group or intervention group. The research team will provide the transportation service to take the participants to the facilities. To guarantee the physical safety of the people who participate, there will be a person certified in life support, who will ensure that the participant who requires entering in the most efficient way to the health system. It is worth clarifying that all study participants will have affiliation to a Health Promoting Entity through which they attend their oncology controls, and additionally, the research group will have a medical insurance policy for the patients who participate in the intervention to cover any event that may arise during it.
3. Collection of qualitative information through focus groups led by an anthropology professional to explore what breast cancer survivors look for in a physical activity program and the main motivations and barriers to attending said program and its acceptability. In addition, information will be collected through interviews with experts who work in health promotion, disease prevention, and cancer patient management to identify those factors that are important to be able to articulate the recreation sector with the health sector in the implementation of a targeted physical activity program for breast cancer survivors. Approximately 10 to 15 interviews will be carried out according to the saturation of the information; the recruitment of these experts will be done through snowball sampling where an expert will refer to contacts related to this topic.

Statistical analyzes will be carried out with SPSS and SAS, an ANOVA analysis of variance, Kruskal-Wallis and McNemar's tests of repeated measures will be carried out to establish the change in the results before and after the intervention. To support the analysis of qualitative data from both the focus groups and the interviews, the NVIVO12 software will be used.

Participants will receive the aggregated results of the general study ensuring confidentiality. Additionally, the participants will receive individually the results of the anthropometric tests and stress tests so that they know their physical condition; those who find a level of risk of coronary heart disease will be explicitly suggested to consult a specialist doctor through their insurer.

ELIGIBILITY:
Inclusion Criteria:

* BCS at least six months post treatment completion
* More than 18 years of age
* Living in Bogotá
* Willing to attend the program and the assessments

Exclusion Criteria:

* The presence of metastatic disease and other health conditions for which community physical activity was contraindicated

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Change in participants' physical activity levels | Physical activity levels were assessed at baseline and after the 8th week
  To assess the change from baseline participants' physical activity levels at 8 weeks, participants wore accelerometers for 7 consecutive days from awakening to bedtime using an elasticized belt around the waist at the right mid-axillary line. For wear-time validation, a minimum of four weekdays and a weekend day with at least 10 hours of wear during the waking time was required. Accelerometers were initialized to collect data at a sampling frequency of 80 Hz, downloaded in one-second epochs and grouped in 60-second epochs for analysis.
Change in participants' motivation to engage in physical activity | Motivational regulation for physical activity was assessed at baseline and after the 8th week
  To assess the change from baseline participants´ motivational regulation for physical activity at 8 weeks, we used the validated Spanish version of the Behavioral Regulation in Exercise Questionnaire-3 [BREQ-3], a 23-item inventory assessing the Self-Determination Theory relevant constructs (which conceptualizes motivation as a continuum ranging from amotivation to a high level of intrinsic motivation). Responses to each item were reported on a 5-point scale ranging from 0 (not true for me) to 4 (very true for me).
Change in participants' quality of life | Quality of life was assessed at baseline and after the 8th week
  To assess the change of quality of life, we used the official Colombian Spanish translation of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire. It incorporates five functioning subscales, three symptom subscales, six single symptoms, an item for illness-related financial difficulties, and a two-item general health/global QoL subscale. Each item was reported on a 4-point scale ranging from 1 (not at all) to 4 (very much), except for the general health subscale, which response options range from 1 (very poor) to 7 (excellent). High scores on the functioning subscales and the global health status/QoL subscale represent higher quality of life, while high scores on the symptom subscales indicate high levels of symptomatology. We also used a subscale of the EORTC questionnaire specific to breast cancer patients regarding physical symptoms for lymphedema; it comprises seven items with responses also ranging from 1 (not at all) to 4 (very much).
Acceptability of My Body | Semi-structured interviews were conducted after the 8th week
  We used a semi-structured interviewing technique to ensure in-depth insights about BCS' perspectives towards physical activity, their anticipated and actual experienced barriers and facilitators to engage in the physical activity intervention, their expected and reported benefits from the physical activity intervention, and the perceived positive and negative aspects of the program.

SECONDARY OUTCOMES:
Sociodemographic variables | Surveys were collected at the baseline
  To characterize the population, we collected surveys inquiring about sociodemographic variables (i.e., age, education, socioeconomic level, employment status, healthcare access).
Body mass index | BMI was assessed at the baseline
  Anthropometric data (height, weight) were directly measured by trained interviewers according to standardized procedures using scale and stadiometer. Body mass index (BMI) was calculated using the formula weight (kg)/height2 (m2); and classified according to the World Health Organization BMI classification

CONTACTS AND LOCATIONS:
Overall Officials: Olga Lucía Sarmiento, PhD, Principal Investigator — Department of Public Health, School of Medicine, Universidad de los Andes, Bogotá, Colombia
Locations (1):
- School of Medicine, Universidad de los Andes, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2017 Causes of Death Collaborators. Global, regional, and national age-sex-specific mortality for 282 causes of death in 195 countries and territories, 1980-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1736-1788. doi: 10.1016/S0140-6736(18)32203-7. Epub 2018 Nov 8. PMID 30496103
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Pardo Ramos C, Cendales Duarte R. Incidencia, Mortalidad y Prevalencia de Cáncer En Colombia 2007-2011.; 2011.
- [Background] María Isabel Calderón Cortés, Ospino MCO, Gianna María Henriquez Mendoza, Molina CÁ. Boletín legislativo & político. Salud Pública del Inst Nac Cancerol. Published online 2018:23.
- [Background] Allemani C, Matsuda T, Di Carlo V, Harewood R, Matz M, Niksic M, Bonaventure A, Valkov M, Johnson CJ, Esteve J, Ogunbiyi OJ, Azevedo E Silva G, Chen WQ, Eser S, Engholm G, Stiller CA, Monnereau A, Woods RR, Visser O, Lim GH, Aitken J, Weir HK, Coleman MP; CONCORD Working Group. Global surveillance of trends in cancer survival 2000-14 (CONCORD-3): analysis of individual records for 37 513 025 patients diagnosed with one of 18 cancers from 322 population-based registries in 71 countries. Lancet. 2018 Mar 17;391(10125):1023-1075. doi: 10.1016/S0140-6736(17)33326-3. Epub 2018 Jan 31. PMID 29395269
- [Background] Battaglini CL, Mills RC, Phillips BL, Lee JT, Story CE, Nascimento MG, Hackney AC. Twenty-five years of research on the effects of exercise training in breast cancer survivors: A systematic review of the literature. World J Clin Oncol. 2014 May 10;5(2):177-90. doi: 10.5306/wjco.v5.i2.177. PMID 24829866
- [Background] Basen-Engquist K, Alfano CM, Maitin-Shepard M, Thomson CA, Schmitz KH, Pinto BM, Stein K, Zucker DS, Syrjala KL, Fallon E, Doyle C, Demark-Wahnefried W. Agenda for Translating Physical Activity, Nutrition, and Weight Management Interventions for Cancer Survivors into Clinical and Community Practice. Obesity (Silver Spring). 2017 Nov;25 Suppl 2(Suppl 2):S9-S22. doi: 10.1002/oby.22031. PMID 29086526
- [Background] Thompson PD, Arena R, Riebe D, Pescatello LS; American College of Sports Medicine. ACSM's new preparticipation health screening recommendations from ACSM's guidelines for exercise testing and prescription, ninth edition. Curr Sports Med Rep. 2013 Jul-Aug;12(4):215-7. doi: 10.1249/JSR.0b013e31829a68cf. No abstract available. PMID 23851406
- [Background] Department of Health & Human Services. 2018 Physical Activity Guidelines Advisory Committee Scientific Report.; 2018.
- [Background] Mason C, Alfano CM, Smith AW, Wang CY, Neuhouser ML, Duggan C, Bernstein L, Baumgartner KB, Baumgartner RN, Ballard-Barbash R, McTiernan A. Long-term physical activity trends in breast cancer survivors. Cancer Epidemiol Biomarkers Prev. 2013 Jun;22(6):1153-61. doi: 10.1158/1055-9965.EPI-13-0141. Epub 2013 Apr 10. PMID 23576689
- [Background] Underwood JM, Townsend JS, Stewart SL, Buchannan N, Ekwueme DU, Hawkins NA, Li J, Peaker B, Pollack LA, Richards TB, Rim SH, Rohan EA, Sabatino SA, Smith JL, Tai E, Townsend GA, White A, Fairley TL; Division of Cancer Prevention and Control, National Center for Chronic Disease Prevention and Health Promotion, Centers for Disease Control and Prevention (CDC). Surveillance of demographic characteristics and health behaviors among adult cancer survivors--Behavioral Risk Factor Surveillance System, United States, 2009. MMWR Surveill Summ. 2012 Jan 20;61(1):1-23. PMID 22258477
- [Background] Fong AJ, Jones JM, Faulkner G, Sabiston CM. Exploring cancer centres for physical activity and sedentary behaviour support for breast cancer survivors. Curr Oncol. 2018 Oct;25(5):e365-e372. doi: 10.3747/co.25.3858. Epub 2018 Oct 31. PMID 30464686
- [Background] Coletta AM, Marquez G, Thomas P, Thoman W, Bevers T, Brewster AM, Hawk E, Basen-Engquist K, Gilchrist SC. Clinical factors associated with adherence to aerobic and resistance physical activity guidelines among cancer prevention patients and survivors. PLoS One. 2019 Aug 1;14(8):e0220814. doi: 10.1371/journal.pone.0220814. eCollection 2019. PMID 31369653
- [Background] Ministerio de Salud. RESUMEN EJECUTIVO Primeros resultados de la Encuesta Nacional de la Situación Nutricional en Colombia ENSIN - 2015. Published online 2015:64. http://www.ensin.gov.co/Documents/Resumen-ejecutivo-ENSIN-2015.pdf
- [Background] Finne E, Glausch M, Exner AK, Sauzet O, Stolzel F, Seidel N. Behavior change techniques for increasing physical activity in cancer survivors: a systematic review and meta-analysis of randomized controlled trials. Cancer Manag Res. 2018 Oct 30;10:5125-5143. doi: 10.2147/CMAR.S170064. eCollection 2018. PMID 30464612
- [Background] Daley AJ, Crank H, Saxton JM, Mutrie N, Coleman R, Roalfe A. Randomized trial of exercise therapy in women treated for breast cancer. J Clin Oncol. 2007 May 1;25(13):1713-21. doi: 10.1200/JCO.2006.09.5083. PMID 17470863
- [Background] Rogers LQ, Hopkins-Price P, Vicari S, Pamenter R, Courneya KS, Markwell S, Verhulst S, Hoelzer K, Naritoku C, Jones L, Dunnington G, Lanzotti V, Wynstra J, Shah L, Edson B, Graff A, Lowy M. A randomized trial to increase physical activity in breast cancer survivors. Med Sci Sports Exerc. 2009 Apr;41(4):935-46. doi: 10.1249/MSS.0b013e31818e0e1b. PMID 19276838
- [Background] Pinto BM, Ciccolo JT. Physical activity motivation and cancer survivorship. Recent Results Cancer Res. 2011;186:367-87. doi: 10.1007/978-3-642-04231-7_16. PMID 21113773
- [Background] Grimmett C, Corbett T, Brunet J, Shepherd J, Pinto BM, May CR, Foster C. Systematic review and meta-analysis of maintenance of physical activity behaviour change in cancer survivors. Int J Behav Nutr Phys Act. 2019 Apr 27;16(1):37. doi: 10.1186/s12966-019-0787-4. PMID 31029140
- [Background] Short CE, James EL, Stacey F, Plotnikoff RC. A qualitative synthesis of trials promoting physical activity behaviour change among post-treatment breast cancer survivors. J Cancer Surviv. 2013 Dec;7(4):570-81. doi: 10.1007/s11764-013-0296-4. Epub 2013 Jul 26. PMID 23888337
- [Background] McEwan D, Rhodes RE, Beauchamp MR. What Happens When the Party is Over?: Sustaining Physical Activity Behaviors after Intervention Cessation. Behav Med. 2022 Jan-Mar;48(1):1-9. doi: 10.1080/08964289.2020.1750335. Epub 2020 Apr 10. PMID 32275199
- [Background] Carey RN, Connell LE, Johnston M, Rothman AJ, de Bruin M, Kelly MP, Michie S. Behavior Change Techniques and Their Mechanisms of Action: A Synthesis of Links Described in Published Intervention Literature. Ann Behav Med. 2019 Jul 17;53(8):693-707. doi: 10.1093/abm/kay078. PMID 30304386
- [Background] Brunet J, Burke SM, Sabiston CM. The benefits of being self-determined in promoting physical activity and affective well-being among women recently treated for breast cancer. Psychooncology. 2013 Oct;22(10):2245-52. doi: 10.1002/pon.3287. Epub 2013 Apr 18. PMID 23596106
- [Background] Emslie C, Whyte F, Campbell A, Mutrie N, Lee L, Ritchie D, Kearney N. 'I wouldn't have been interested in just sitting round a table talking about cancer'; exploring the experiences of women with breast cancer in a group exercise trial. Health Educ Res. 2007 Dec;22(6):827-38. doi: 10.1093/her/cyl159. Epub 2007 Jan 31. PMID 17272293
- [Background] Midtgaard J, Rossell K, Christensen JF, Uth J, Adamsen L, Rorth M. Demonstration and manifestation of self-determination and illness resistance--a qualitative study of long-term maintenance of physical activity in posttreatment cancer survivors. Support Care Cancer. 2012 Sep;20(9):1999-2008. doi: 10.1007/s00520-011-1304-8. Epub 2011 Nov 15. PMID 22083498
- [Background] Spector D, Battaglini C, Alsobrooks A, Owen J, Groff D. Do breast cancer survivors increase their physical activity and enhance their health-related quality of life after attending community-based wellness workshops? J Cancer Educ. 2012 Jun;27(2):353-61. doi: 10.1007/s13187-011-0306-z. PMID 22210191
- [Background] Errico KM, Rowden D. Experiences of breast cancer survivor-advocates and advocates in countries with limited resources: a shared journey in breast cancer advocacy. Breast J. 2006 Jan-Feb;12 Suppl 1:S111-6. doi: 10.1111/j.1075-122X.2006.00208.x. PMID 16430394
- [Background] Johnson CM, Molina Y, Blas M, Erickson M, Bayer A, Gutierrez MC, Nevin PE, Alva I, Rao D. "The disease is mine, the body is mine, I decide": Individual, interpersonal, and institutional barriers and facilitators among survivors of women's cancers in Andean countries. Health Care Women Int. 2018 May;39(5):522-535. doi: 10.1080/07399332.2017.1421198. Epub 2018 Feb 2. PMID 29313760
- [Background] Wurz A, St-Aubin A, Brunet J. Breast cancer survivors' barriers and motives for participating in a group-based physical activity program offered in the community. Support Care Cancer. 2015 Aug;23(8):2407-16. doi: 10.1007/s00520-014-2596-2. Epub 2015 Jan 22. PMID 25605568
- [Background] Sabiston CM, Fong AJ, O'Loughlin EK, Meterissian S. A mixed-methods evaluation of a community physical activity program for breast cancer survivors. J Transl Med. 2019 Jun 19;17(1):206. doi: 10.1186/s12967-019-1958-4. PMID 31217021
- [Background] Diaz Del Castillo A, Gonzalez SA, Rios AP, Paez DC, Torres A, Diaz MP, Pratt M, Sarmiento OL. Start small, dream big: Experiences of physical activity in public spaces in Colombia. Prev Med. 2017 Oct;103S:S41-S50. doi: 10.1016/j.ypmed.2016.08.028. Epub 2016 Aug 26. PMID 27575321
- [Background] Torres A, Diaz MP, Hayat MJ, Lyn R, Pratt M, Salvo D, Sarmiento OL. Assessing the effect of physical activity classes in public spaces on leisure-time physical activity: "Al Ritmo de las Comunidades" A natural experiment in Bogota, Colombia. Prev Med. 2017 Oct;103S:S51-S58. doi: 10.1016/j.ypmed.2016.11.005. Epub 2016 Nov 12. PMID 27847217
- [Background] Boing L, Baptista F, Pereira GS, Sperandio FF, Moratelli J, Cardoso AA, Borgatto AF, de Azevedo Guimaraes AC. Benefits of belly dance on quality of life, fatigue, and depressive symptoms in women with breast cancer - A pilot study of a non-randomised clinical trial. J Bodyw Mov Ther. 2018 Apr;22(2):460-466. doi: 10.1016/j.jbmt.2017.10.003. Epub 2017 Oct 12. PMID 29861250
- [Background] Schmidt T, Rudolph I, Wozniak T, Ruetters D, Van Mackelenbergh MT, Huebner J. Effect of ballroom dancing on the well-being of cancer patients: Report of a pilot project. Mol Clin Oncol. 2018 Sep;9(3):342-346. doi: 10.3892/mco.2018.1663. Epub 2018 Jun 28. PMID 30112180
- [Background] World Economic Forum. The Inclusive Development Index 2018 Summary and Data Highlights.; 2018.
- [Background] Gaffney LK, Lozano OD, Almanza A, Ruiz N, Mantero A, Stoutenberg M. The Implementation of a National Physical Activity Intervention in Colombia. J Phys Act Health. 2019 Jun 1;16(6):430-436. doi: 10.1123/jpah.2018-0183. Epub 2019 May 19. PMID 31104541
- [Background] Pluye P, Hong QN. Combining the power of stories and the power of numbers: mixed methods research and mixed studies reviews. Annu Rev Public Health. 2014;35:29-45. doi: 10.1146/annurev-publhealth-032013-182440. Epub 2013 Oct 30. PMID 24188053
- [Background] Pudkasam S, Polman R, Pitcher M, Fisher M, Chinlumprasert N, Stojanovska L, Apostolopoulos V. Physical activity and breast cancer survivors: Importance of adherence, motivational interviewing and psychological health. Maturitas. 2018 Oct;116:66-72. doi: 10.1016/j.maturitas.2018.07.010. Epub 2018 Jul 23. PMID 30244781
- [Background] Karageorghis CI, Jones L, Priest DL, Akers RI, Clarke A, Perry JM, Reddick BT, Bishop DT, Lim HB. Revisiting the relationship between exercise heart rate and music tempo preference. Res Q Exerc Sport. 2011 Jun;82(2):274-84. doi: 10.1080/02701367.2011.10599755. PMID 21699107
- [Background] Yamashita S, Iwai K, Akimoto T, Sugawara J, Kono I. Effects of music during exercise on RPE, heart rate and the autonomic nervous system. J Sports Med Phys Fitness. 2006 Sep;46(3):425-30. PMID 16998447
- [Background] Freedson PS, Melanson E, Sirard J. Calibration of the Computer Science and Applications, Inc. accelerometer. Med Sci Sports Exerc. 1998 May;30(5):777-81. doi: 10.1097/00005768-199805000-00021. PMID 9588623
- [Background] Teixeira PJ, Carraca EV, Markland D, Silva MN, Ryan RM. Exercise, physical activity, and self-determination theory: a systematic review. Int J Behav Nutr Phys Act. 2012 Jun 22;9:78. doi: 10.1186/1479-5868-9-78. PMID 22726453
- [Background] Gonzalez-Cutre D, Sicilia A, Fernandez A. [Toward a deeper understanding of motivation towards exercise: measurement of integrated regulation in the Spanish context]. Psicothema. 2010 Nov;22(4):841-7. Spanish. PMID 21044522
- [Background] Finck C, Barradas S, Zenger M, Hinz A. Quality of life in breast cancer patients: Associations with optimism and social support. Int J Clin Health Psychol. 2018 Jan-Apr;18(1):27-34. doi: 10.1016/j.ijchp.2017.11.002. Epub 2017 Dec 9. PMID 30487907
- [Background] Finck C, Barradas S, Singer S, Zenger M, Hinz A. Health-related quality of life in Colombia: reference values of the EORTC QLQ-C30. Eur J Cancer Care (Engl). 2012 Nov;21(6):829-36. doi: 10.1111/ecc.12000. Epub 2012 Sep 12. PMID 22966808
- [Background] Sallis JF, Cervero RB, Ascher W, Henderson KA, Kraft MK, Kerr J. An ecological approach to creating active living communities. Annu Rev Public Health. 2006;27:297-322. doi: 10.1146/annurev.publhealth.27.021405.102100. PMID 16533119
- [Background] Wirtz P, Baumann FT. Physical Activity, Exercise and Breast Cancer - What Is the Evidence for Rehabilitation, Aftercare, and Survival? A Review. Breast Care (Basel). 2018 Apr;13(2):93-101. doi: 10.1159/000488717. Epub 2018 Apr 11. PMID 29887785
- [Background] Rogers LQ, Vicari S, Courneya KS. Lessons learned in the trenches: facilitating exercise adherence among breast cancer survivors in a group setting. Cancer Nurs. 2010 Nov-Dec;33(6):E10-7. doi: 10.1097/NCC.0b013e3181db699d. PMID 20562618
- [Background] Cerulli C, Parisi A, Sacchetti M, et al. Dancing with health: A new dance protocol to improve the quality of life of breast cancer survivors. Med dello Sport. 2019;72(2):295-304. doi:10.23736/S0025-7826.19.03530-0
- [Background] Leach HJ, Danyluk JM, Culos-Reed SN. Design and implementation of a community-based exercise program for breast cancer patients. Curr Oncol. 2014 Oct;21(5):267-71. doi: 10.3747/co.21.2079. PMID 25302035
- [Background] Caperchione CM, Sabiston CM, Stolp S, Bottorff JL, Campbell KL, Eves ND, Ellard SL, Gotay C, Sharp P, Pullen T, Fitzpatrick KM. A preliminary trial examining a 'real world' approach for increasing physical activity among breast cancer survivors: findings from project MOVE. BMC Cancer. 2019 Mar 27;19(1):272. doi: 10.1186/s12885-019-5470-2. PMID 30917793
- [Background] Szalai M, Szirmai A, Fuge K, Makai A, Erdelyi G, Premusz V, Bodis J. Special aspects of social support: Qualitative analysis of oncologic rehabilitation through a belly dancing peer support group. Eur J Cancer Care (Engl). 2017 Nov;26(6). doi: 10.1111/ecc.12656. Epub 2017 Feb 13. PMID 28194904
- [Background] Balneaves LG, Van Patten C, Truant TL, Kelly MT, Neil SE, Campbell KL. Breast cancer survivors' perspectives on a weight loss and physical activity lifestyle intervention. Support Care Cancer. 2014 Aug;22(8):2057-65. doi: 10.1007/s00520-014-2185-4. Epub 2014 Mar 15. PMID 24633590
- [Background] Loh SY, Chew SL, Lee SY. Physical activity and women with breast cancer: insights from expert patients. Asian Pac J Cancer Prev. 2011;12(1):87-94. PMID 21517237
- [Result] Obesity: preventing and managing the global epidemic. Report of a WHO consultation. World Health Organ Tech Rep Ser. 2000;894:i-xii, 1-253. PMID 11234459
- [Derived] Rubio MA, Mejia-Arbelaez CM, Wilches-Mogollon MA, Moreno S, Finck C, Rosas LG, Romero SA, Guevara P, Cabas S, Rubiano O, Florez-Pregonero A, Leon JG, Alarcon LF, Haile R, Sarmiento OL, King AC. "My Body, My Rhythm, My Voice": a community dance pilot intervention engaging breast cancer survivors in physical activity in a middle-income country. Pilot Feasibility Stud. 2023 Feb 28;9(1):30. doi: 10.1186/s40814-023-01253-x. PMID 36855214

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT05252780/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT05252780/ICF_001.pdf